CLINICAL TRIAL: NCT01202266
Title: A Phase 1 Placebo-Controlled Study To Assess The Safety, Tolerability And Pharmacokinetics Of Pf-05161704 After Administration Of Multiple Escalating Oral Doses In Healthy Volunteers
Brief Title: A Multiple Dose Study Of PF-05161704 In Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated on October 29, 2010 due to gastrointestinal adverse events.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B2911002
Record Dates: First submitted 2010-09-13; First posted 2010-09-15 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Multiple Ascending Dose; Phase 1; Safety and Tolerability; PK; Healthy Subjects
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- 5 mg PF-05161704 or Placebo (Experimental)
  Interventions: Drug: PF-05161704 or Placebo
- 15 mg PF-05161704 or Placebo (Experimental): Planned dose: may be modified based on emerging PK and safety data.
  Interventions: Drug: PF-05161704 or Placebo
- 50 mg PF-05161704 or Placebo (Experimental): Planned dose: may be modified based on emerging PK and safety data.
  Interventions: Drug: PF-05161704 or Placebo
- 150 mg PF-05161704 or Placebo (Experimental): Planned dose: may be modified based on emerging PK and safety data.
  Interventions: Drug: PF-05161704 or Placebo
- xx mg PF-05161704 or Placebo (Experimental): Planned dose and dosing regimen will be determined based on emerging PK and safety data.
  Interventions: Drug: PF-05161704 or Placebo
- xxx mg PF-05161704 or Placebo (Experimental): Dose will be determined based on data from previous 5 arms.
  Interventions: Drug: PF-05161704 or Placebo
- yy mg PF-05161704 or Placebo (Experimental): Dose will be determined based on data from previous 6 arms
  Interventions: Drug: PF-05161704 or Placebo
- yyy mg PF-05161704 or Placebo (Experimental): Dose will be determined based on data from previous 7 arms.
  Interventions: Drug: PF-05161704 or Placebo

INTERVENTIONS:
Drug: PF-05161704 or Placebo — PF-05161704 and Placebo (3:1) oral dosing Suspensions administered twice daily for 14 days immediately after breakfast and dinner
  Arms: 5 mg PF-05161704 or Placebo
Drug: PF-05161704 or Placebo — PF-05161704 and Placebo (3:1) oral dosing Suspensions administered twice daily for 14 days immediately after breakfast and dinner
  Arms: 15 mg PF-05161704 or Placebo
Drug: PF-05161704 or Placebo — PF-05161704 and Placebo (3:1) oral dosing Suspensions administered twice daily for 14 days immediately after breakfast and dinner
  Arms: 50 mg PF-05161704 or Placebo
Drug: PF-05161704 or Placebo — PF-05161704 and Placebo (3:1) oral dosing Suspensions administered twice daily for 14 days immediately after breakfast and dinner
  Arms: 150 mg PF-05161704 or Placebo
Drug: PF-05161704 or Placebo — PF-05161704 and Placebo (3:1) oral dosing Suspensions administered twice daily for 14 days immediately after breakfast and dinner or once daily for 14 days immediately after breakfast
  Arms: xx mg PF-05161704 or Placebo
Drug: PF-05161704 or Placebo — PF-05161704 and Placebo (3:1) oral dosing Suspensions administered once daily for 14 days immediately after breakfast
  Arms: xxx mg PF-05161704 or Placebo
Drug: PF-05161704 or Placebo — PF-05161704 and Placebo (3:1) oral dosing Suspensions administered once daily for 14 days immediately after breakfast
  Arms: yy mg PF-05161704 or Placebo
Drug: PF-05161704 or Placebo — PF-05161704 and Placebo (3:1) oral dosing Suspensions administered once daily for 14 days immediately after breakfast
  Arms: yyy mg PF-05161704 or Placebo

SUMMARY:
The primary purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of multiple escalating oral doses of PF-05161704 in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female (non-childbearing potential) subjects between the ages of 18 and 55 years, inclusive
* Body Mass Index (BMI) of 24.5 to 35.5 kg/m2 and a total body weight >50 kg (110 lbs.)

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (e.g., gastrectomy).
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
* History or evidence of habitual use of tobacco or nicotine containing products within 3 months of screening or positive cotinine test at screening or Day -1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability endpoints evaluated by adverse event monitoring, laboratory values, cardiovascular monitoring | 2 weeks
Pharmacokinetic Endpoints: single dose and steady state pharmacokinetics of PF-05161704 and its metabolite PF-05200145. Urinary recovery will also be assessed for PF-05161704 and PF-05200145 | 2 weeks

SECONDARY OUTCOMES:
Pharmacodynamic Endpoints: Absolute value and change from Day 0 baseline in postprandial GLP-1. Postprandial plasma PYY, triglycerides and apoB48. Absolute value and change from baseline in apoB100 and VLDL | 2 weeks
Exploratory Parameters: absolute value and change from Day 0 baseline in concentrations of fasting serum lipids and body weight | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2911002&StudyName=A%20Multiple%20Dose%20Study%20Of%20PF-05161704%20In%20Healthy%20Volunteers